CLINICAL TRIAL: NCT01622855
Title: Prevention of Post-Rape Psychopathology and Drug Abuse
Brief Title: Acute Intervention to Reduce Distress Following Sexual Assault
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCT11158; R01DA011158 (NIH)
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Drug Use; Drug Abuse; Posttraumatic Stress Disorder
Keywords: Rape; Secondary prevention; Intervention
MeSH Terms: conditions — Substance-Related Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PPRS video (Experimental): Prevention of post sexual assault stress
  Interventions: Behavioral: PPRS
- Standard care (No Intervention): Receipt of standard services

INTERVENTIONS:
Behavioral: PPRS — Video including psycho-education and modeling of adaptive behavioral coping strategies for use post-assault.
  Arms: PPRS video

SUMMARY:
The purpose of this study was to evaluate whether a brief intervention in video format delivered in the post assault medical exam setting and including education about assault reactions and instruction in and modeling of successful coping strategies would reduce post assault drug use or abuse and PTSD symptoms as compared to standard care.

DETAILED DESCRIPTION:
The intervention being evaluated was shown at the time of the post assault medical exam and includes two main components: preparation for the medical exam; and information about and modelling of coping strategies that may help women cope in the aftermath of assault. The intervention content is delivered via video. Intervention and standard care groups were compared with regard to measures of substance use and abuse and symptoms of PTSD and other potentially comorbid problems including symptoms of depression or other anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Seeking medical care after recent sexual assault

Exclusion Criteria:

* Active psychosis
* Active suicidality
* Cognitive impairment
* Non-English speaking
* Severe injury

Ages: 14 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 1997-03; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Frequency of specific drug use | 14 days
  Number of days use of specific drugs in preceding 14 days at 6 week, 3 and 6 month follow-ups

SECONDARY OUTCOMES:
Specific Drug Abuse | 1.5, 3, 6 months
  Criteria for DSM-IV substance abuse based on structured interview
PSS-SR | 2 weeks
  Measure of PTSD symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Resnick, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States